CLINICAL TRIAL: NCT02814955
Title: Study of Electrophysiological Effects of NACOS and AVK on the Pulmonary Veins and the Left Atrium of Patients Referred for Paroxysmal AF Catheter Ablation
Brief Title: Electrophysiological Effects of NACOS and AVK on Pulmonary Veins and Left Atrium in Paroxysmal AF Catheter Ablation
Acronym: NACO-VP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A15-D20-VOL.25
Record Dates: First submitted 2016-06-15; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pulmonary veins; oral anticoagulant; electrophysiology; anticoagulant drugs
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — cordarone
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- referred for paroxysmal atrial fibrillation with fluindione
- referred for paroxysmal atrial fibrillation with previscan
- referred for paroxysmal atrial fibrillation with apixaban
- referred for paroxysmal atrial fibrillation with rivaroxaban
- referred for paroxysmal atrial fibrillation with dabigatran

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmias with a constantly growing prevalence AF. The purpose of paroxysmal AF processing is to control outbreaks from these pulmonary veins, medicated way (antiarrhythmic) or interventional. Ablation (radiofrequency or cryotherapy) has become in this context recognized and effective treatment of AF. In addition, antithrombotic treatments in this context is a major treatments for the prevention of stroke (stroke). They are most often associated with antiarrhythmic treatment to prevent recurrence of AF or to slow it during a relapse.

Recent experimental studies have highlighted the direct electrophysiological properties of dabigatran and rivaroxaban in the pulmonary veins and the left atrium. Dabigatran demonstrated in this study that it induced a prolongation of potential action in the pulmonary veins and the left atrium and it decreased the incidence of FA-induced by stimulation. Conversely, rivaroxaban induces shortening of the action potential in the left atrium (untested properties in the pulmonary veins). To our knowledge, apixaban and warfarin have not been studied in this context.

It is therefore possible that some of the new oral anticoagulants (NACOS) or some AVK (fluindione and warfarin), have direct electrophysiological effects in the pulmonary veins and on the left atrium and could influence AF recurrences (with effect " antiarrhythmic-like "or rather a pro-arrhythmic effect) after ablation.A retrospective analysis conducted at the University Hospital of Caen on very low numbers suggest that patients on dabigatran would have less pulmonary veins connected in early ablation procedure that patients on warfarin or rivaroxaban. Despite the limitations inherent in this analysis (very low numbers, retrospective analysis, unique setting and having studied his own limits), these results are consistent with the fundamental studies, and thus encourage us to pursue our hypothesis to obtain more statistical power and reliability in our measurements and results.

We therefore propose the study of the electrophysiological effects of NACOS (apixaban, dabigatran, rivaroxaban) and warfarin (warfarin and fluindione) on the pulmonary veins and the left atrium of patients referred for ablation of paroxysmal AF (radiofrequency or cryotherapy ) the CHU of Caen and Tours and clinic Saint Martin Caen.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients for ablation of paroxysmal AF
* On healthy heart
* Sinus rhythm during the procedure
* Patient> 18 years

Exclusion Criteria:

* Patient <18 years
* Severe Mitral valve disease,
* underlying heart disease
* Patients refusing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to all patients referred for paroxysmal atrial fibrillation radiofrequency ablation , clinically stable, at Caen University Hospital, Tours and Saint-Martin clinic.
  These patients have a strict, rigorous and systematic follow after these ablation at 1, 3 and 6 months with routine ECG.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Reccurence of atrial fibrillation | 6 months

SECONDARY OUTCOMES:
number of active pulmonary veins | 1 day
  Measure at the ostia with the lasso
Spontaneous cycle length in active pulmonary veins | 1 day
  Measure at the ostia with the lasso
Number of connected pulmonary veins | 1 day
  Measure at the ostia with the lasso
Measure of refractory period for each pulmonary veins and left atria | 1 day
  Measure at the ostia with the lasso for each VP, and with coronary sinus for the LA.
Number of re-connected pulmonary veins with ATP | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: Yes